CLINICAL TRIAL: NCT01290107
Title: MLL Rearrangements in Acute Myeloid Leukemia: A Pilot Project to Expand and Study MLL-ENL in NOD SCID Gamma Mice
Brief Title: Biomarkers in Samples of Bone Marrow From Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML11B7; COG-AAML11B7 (Other: Children's Oncology Group); NCI-2011-02847 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AAML11B7 (Other: Children's Oncology Group)
Record Dates: First submitted 2011-02-03; First posted 2011-02-04 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; childhood acute myeloid leukemia/other myeloid malignancies
MeSH Terms: conditions — Leukemia; Congenital Abnormalities | interventions — Gene Rearrangement; Microarray Analysis; Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone Marrow
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA analysis
Genetic: gene rearrangement analysis
Genetic: microarray analysis
Genetic: polymerase chain reaction
Other: immunological diagnostic method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of bone marrow from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is looking at bone marrow samples from patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To successfully transplant human acute myeloid leukemia (AML) cells into immunocompromised mice for the purpose of expansion of the cells.
* To harvest the cells and use chromatin immunoprecipitation (ChIP) methods to identify the locations of the protein complexes on the genome.
* To study the interactions of the Super Elongation Complex (SEC) and Dot1 Complex (DotCom) complexes in human leukemia samples.
* To compare the genomic targets of the complexes formed by MLL-ENL chimeras to non-MLL-rearranged leukemia samples to normal controls.

OUTLINE: Cryopreserved cells are implanted into NOD SCID gamma mice, expanded, harvested, and studied by chromatin immunoprecipitation (ChIP) methods (using antibodies to ENL, Af9, and AF10). Results are then analyzed by PCR, DNA sequencing, and/or microarray analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia (AML)
* Cryopreserved mixed-lineage leukemia (MLL) ENL AML rearrangement cells, normal karyotype and non-MLL rearrangement AML cells, and non-leukemic bone marrow samples from the COG tissue bank

  * 3 specimens of each type

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosis of acute myeloid leukemia.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Estimated)
Dates: Start 2011-02; Primary Completion 2015-01 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Successful transplantation of human acute myeloid leukemia (AML) cells into immunocompromised mice for the purpose of expansion of the cells

SECONDARY OUTCOMES:
Identification of the locations of the protein complexes
Interactions of the SEC and DotCom complexes in human leukemia samples

CONTACTS AND LOCATIONS:
Overall Officials: Eric Guest, MD, Principal Investigator — Children's Mercy Hospital Kansas City